CLINICAL TRIAL: NCT01873092
Title: AMBULATORY OXIMETRY MONITORING (AOM): a New Approach to Quantify Oxygen Desaturation in Ambulatory COPD Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Miriam D Cohen, Nurse Practitioner, VA New York Harbor Healthcare System
Other Study IDs: 00493
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Oximetry; Physical Activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with COPD: Patients who meet criteria for chronic obstructive pulmonary disease

SUMMARY:
Chronic obstructive lung disease (COPD) is characterized by airflow obstruction that is progressive over many years and is largely irreversible. Advanced COPD is associated with arterial oxygen desaturation leading to a series of complications and, ultimately, decreased survival. Long-term oxygen therapy can improve clinical outcomes in these patients, but the exact target of oxygen saturation that actually translates into improvements is not known. The basis for the work in this proposal is to focus a new approach to measure oxygen desaturation linked to daily activity. Accelerometers are used to measure daily activity and then synchronized with ambulatory oximetry to establish an activity/oxygen-saturation profile for individual patients. The three main objectives of this study are 1) determine the feasibility of AOM as a measurement of the temporal profile of oxygen saturation in patients with chronic lung disease; 2) determine if serial AOM-derived data is reliable and reproducible; and 3) determine thresholds of oxygen desaturation that are associated with different activity profiles

ELIGIBILITY:
Inclusion Criteria:

1. Veteran patients with a diagnosis of COPD or other chronic lung disease
2. able to read and understand English
3. > 45 years old
4. ambulatory and able to perform functional testing

Exclusion Criteria:

1. unable or unwilling to give informed consent
2. daily use of a motorized cart
3. impairment of cognition or communication
4. history of drug or alcohol treatment within the past 6 months
5. poor peripheral blood flow to the finger rendering oxygen saturation by pulse oximetry unreliable
6. Recent acute medical events (chest pain, discomfort, etc) that would suggest a contraindication to participate at the scheduled time

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veteran patients with chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2003-05; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Ambulatory oximetry/activity profile | Data is collected over 30-34 consecutive hours
  Oxygen saturation is measured with a pulse oximeter that has the capacity to collect data over 30- 34 hours; physical activity is measured with two pizo-electric accelerometers. Oximetry and activity data are synchronized to define a profile of oxygen saturation that is linked to usual daily activity.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Cohen, Principal Investigator — VA New York Harbor Healthcare System
Locations (1):
- VA, New York Harbor Healthcare Service, Brooklyn, New York, United States

REFERENCES:
- [Result] Cohen MD, Cutaia M. A novel approach to measuring activity in chronic obstructive pulmonary disease: using 2 activity monitors to classify daily activity. J Cardiopulm Rehabil Prev. 2010 May-Jun;30(3):186-94. doi: 10.1097/HCR.0b013e3181d0c191. PMID 20216326
- [Result] Cohen MD, Cutaia M, Brehm R, Brutus V, Pike VC, Lewendowski D. Detecting motor vehicle travel in accelerometer data. COPD. 2012 Apr;9(2):102-10. doi: 10.3109/15412555.2011.650238. Epub 2012 Mar 12. PMID 22409288
- [Result] Cutaia M, Brehm R, Cohen M. The relationship of the BODE index to oxygen saturation during daily activities in patients with chronic obstructive pulmonary disease. Lung. 2011 Aug;189(4):269-77. doi: 10.1007/s00408-011-9308-1. Epub 2011 Jun 24. PMID 21701832